CLINICAL TRIAL: NCT04352959
Title: COVID-19: Nasal and Salivary Detection of the SARS-CoV-2 Virus After Antiviral Mouthrinses: Double-blind, Randomized, Placebo-controlled Clinical Study
Brief Title: COVID-19: Nasal and Salivary Detection of the SARS-CoV-2 Virus After Antiviral Mouthrinses
Acronym: BBCovid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claude Bernard University (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Carrouel Florence, Associate professor, Claude Bernard University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BBCovid
Record Dates: First submitted 2020-04-15; First posted 2020-04-20 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: COVID19; Mouthwash; Saliva
Keywords: covid19; SARS-CoV-2; mouthrinses; antiviral; bêta-cyclodextrin; citrox
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mouth rinse with antiviral (Active Comparator)
  Interventions: Device: mouthrinse with bêta-cyclodextrin and citrox
- mouth rinse without antiviral (Placebo Comparator)
  Interventions: Device: mouthrinse without bêta-cyclodextrin and citrox

INTERVENTIONS:
Device: mouthrinse with bêta-cyclodextrin and citrox — 3 daily mouthrinses for 7 days
  Arms: mouth rinse with antiviral
Device: mouthrinse without bêta-cyclodextrin and citrox — 3 daily mouthrinses for 7 days
  Arms: mouth rinse without antiviral

SUMMARY:
Given the current lack of effective COVID-19 treatment, it is necessary to explore alternative methods to contain the spread of the infection, focusing in particular on its mode of transmission. The modes of person-to-person transmission of SARS-CoV-2 are direct transmission, such as sneezing, coughing, transmission through inhalation of small droplets, and transmission through contact, such as contact with nasal, oral and eye mucous membranes. SARS-CoV-2 can also be transmitted directly or indirectly through saliva. The use of antiviral mouthrinses may be used as adjunctive therapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Covid-19 infection by the patient's general practitioner and hospital doctor
* Clinical signs started less than 8 days ago.
* Virological confirmation
* Understanding and acceptance of the trial.
* Written agreement to participate in the trial

Exclusion Criteria:

* Pregnancy
* Breastfeeding
* Inability to comply with protocol
* Lack of written agreement

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline amount of SARS-CoV-2 in salivary samples at 7 days | 7 days
  Quantitative PCR experiments will be performed and a quantitative analysis of the salivary samples will be made

SECONDARY OUTCOMES:
Change from Baseline amount of SARS-CoV-2 virus in nasal samples at 7 days | 7 days
  Quantitative PCR experiments will be performed and a quantitative analysis of the nasal samples will be made

CONTACTS AND LOCATIONS:
Overall Officials: Florence Carrouel, Dr, Study Director — University Claude Bernard Lyon 1
Locations (4):
- France (4):
  - Clinic of the Protestant Infirmary in Lyon, Caluire-et-Cuire
  - Hospital Center Emile Roux, Le Puy-en-Velay
  - Hospital Center Saint Luc Saint Joseph, Lyon
  - Intercommunal Hospital Center of Mont de Marsan, Mont-de-Marsan

REFERENCES:
- [Background] Carrouel F, Conte MP, Fisher J, Goncalves LS, Dussart C, Llodra JC, Bourgeois D. COVID-19: A Recommendation to Examine the Effect of Mouthrinses with beta-Cyclodextrin Combined with Citrox in Preventing Infection and Progression. J Clin Med. 2020 Apr 15;9(4):1126. doi: 10.3390/jcm9041126. PMID 32326426
- [Background] Carrouel F, Goncalves LS, Conte MP, Campus G, Fisher J, Fraticelli L, Gadea-Deschamps E, Ottolenghi L, Bourgeois D. Antiviral Activity of Reagents in Mouth Rinses against SARS-CoV-2. J Dent Res. 2021 Feb;100(2):124-132. doi: 10.1177/0022034520967933. Epub 2020 Oct 22. PMID 33089717
- [Derived] Carrouel F, Viennot S, Valette M, Cohen JM, Dussart C, Bourgeois D. Salivary and Nasal Detection of the SARS-CoV-2 Virus After Antiviral Mouthrinses (BBCovid): A structured summary of a study protocol for a randomised controlled trial. Trials. 2020 Nov 2;21(1):906. doi: 10.1186/s13063-020-04846-6. PMID 33138848
- [Derived] Burton MJ, Clarkson JE, Goulao B, Glenny AM, McBain AJ, Schilder AG, Webster KE, Worthington HV. Antimicrobial mouthwashes (gargling) and nasal sprays administered to patients with suspected or confirmed COVID-19 infection to improve patient outcomes and to protect healthcare workers treating them. Cochrane Database Syst Rev. 2020 Sep 16;9(9):CD013627. doi: 10.1002/14651858.CD013627.pub2. PMID 32936948